CLINICAL TRIAL: NCT07344376
Title: An Extension Study to Assess the Long-term Safety and Efficacy of Hunterase (Idursulfase Beta) in Patients With Hunter Syndrome
Brief Title: An Extension Study to Assess the Long-term Safety and Efficacy of Hunterase (Idursulfase Beta)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GC Biopharma Corp (Industry)
Collaborators: Samsung Medical Center, Sungkyunkwan University School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC1111_P3_Ex
Record Dates: First submitted 2025-11-17; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: MPS II; Hunter Syndrome (MPS II); Hunter Syndrome; Hunterase; GC1111
Keywords: Hunterase; GC1111; GC Biopharma; Long-term study; extension study
MeSH Terms: conditions — Sudden Infant Death; Mucopolysaccharidosis II

STUDY DESIGN:
Intervention Model Description: Phase 3 Extension study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hunterase (Other): Single arm
  Interventions: Drug: Hunterase

INTERVENTIONS:
Drug: Hunterase — 0.5mg/kg weekly IV administration
  Other Names: GC1111

SUMMARY:
The objective of this study is to assess the long-term safety and efficacy of Hunterase for approximately 1 year in subjects who completed the end of study (EOS) visit (Visit 54) tests in the Phase 3 Hunterase study and patients who received Hunterase for more than 6 months

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed with Hunter syndrome (MPS II) who completed activities at the EOS visit (Visit 54) in the GC1111_P3 study
2. (Subject who did not participate in the GC1111_P3 study) Subject diagnosed with Hunter syndrome (MPS II) who received Hunterase for more than 6 months
3. (Subjects who did not participate in the GC1111_P3 study) Males aged ≥ 5
4. Informed consent form voluntarily signed by the subject or by a legally acceptable representative
5. Subject who agrees to use contraception

Exclusion Criteria:

1. Subject with hypersensitivity to any of the ingredients of the investigational product
2. Subject impossible to perform follow-up observation of the safety
3. Subject who received the treatment with another investigational product within 14 days prior to the start of study drug
4. Subject who plans to be treated with another investigational product during the study period
5. Subject who has history of tracheostomy, bone marrow transplant, or cord blood transplant
6. Any other inappropriate conditions for study participation at the investigator's discretion

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 30 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Laboratory tests (CBC, Chemistry, Urinanalysis) | Every visit until 12months
  Abnormality of Laboratory tests results
Physical examination | Every visit until 12months
  Abnormality of physical examination
Adverse Event | Every visit until 12months
  occurence, grade
Electrocardiography | Every 6 months until 12months
  Abnormality of ECG results

SECONDARY OUTCOMES:
6-minute walk test | Every 4months until 12months
  Mean, Change and percent change of 6-minute walk test
Urine GAG (Heparan sulfate, Dermatan sulfate) | Every visit until 12months
  Mean, Change and percent change of Urine HS/DS

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No